CLINICAL TRIAL: NCT03673657
Title: A Prospective, Single-arm, Phase II Study of Early Nutritional Intervention During Concurrent Chemoradiotherapy for Local Advanced Non-small Cell Lung Cancer
Brief Title: Study of Early Nutritional Intervention During Concurrent Chemoradiotherapy for Local Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1041
Record Dates: First submitted 2018-09-05; First posted 2018-09-17 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Local Advanced Non-small Cell Lung Cancer
Keywords: Local Advanced Non-small Cell Lung Cancer; Chemoradiotherapy; Early nutritional intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study group (Experimental): Patients in the study group received early nutritional intervention, including individualized nutrition counseling and oral nutritional supplements from the initiation of CCRT to 2 weeks after its completion. Energy goal: daily total nutritional intake of about 30 kcal/kg.
  Definitive thoracic radiotherapy with total radiation doses of 60-68 Gy; Weekly DP chemotherapy concurrent with thoracic radiotherapy.
  Interventions: Dietary Supplement: Early Nutrition Intervention from the start of CCRT; Radiation: Thoracic radiotherapy; Drug: Weekly DP chemotherapy concurrent with thoracic radiotherapy

INTERVENTIONS:
Dietary Supplement: Early Nutrition Intervention from the start of CCRT — Nutrition counseling and oral nutritional supplements from the start of radiotherapy; weekly counseling sessions; daily energy intake of approximately 30 kcal/kg.
Radiation: Thoracic radiotherapy — Definitive thoracic radiotherapy with total radiation doses of 60-68 Gy
Drug: Weekly DP chemotherapy concurrent with thoracic radiotherapy — Weekly docetaxel (25mg/㎡) and nedaplatin (25mg/㎡) concurrent with thoracic radiotherapy

SUMMARY:
This single-arm phase II prospective study is to determine the efficacy of early nutritional intervention during concurrent chemoradiotherapy for local advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This single-arm phase II prospective study is to determine the efficacy of early nutritional intervention during concurrent chemoradiotherapy for local advanced non-small cell lung cancer.

Patients in the study group received early nutritional intervention, including individualized nutrition counseling and oral nutritional supplements from the initiation of CCRT to 2 weeks after its completion. Weekly counseling sessions, conducted by both doctors and nurses, aimed to educate patients on regulating their regular dietary intake to meet specific energy, protein, and other macronutrient requirements. Dietary advice provided precise instructions on food type and quantity, meal frequency, and calorie or protein intake to ensure a daily energy intake of approximately 30 kcal/kg. All patients received definitive thoracic radiotherapy with total radiation doses of 60-68 Gy, concurrent with weekly docetaxel (25mg/㎡) and nedaplatin (25mg/㎡).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed unresectable stage IIIA-IIIC non-small cell lung cancer.
* Recieved definitive concurrent chemoradiotherapy.
* Pretreatment PG-SGA score A or B.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Estimated life expectancy of at least 6 months.
* Without contraindication for chemoradiotherapy.

Exclusion Criteria:

* Severe impairment of intestinal function, or intolerance of enteral nutrition.
* Severe vomiting, gastrointestinal bleeding, or intestinal obstruction.
* Severe malnutrition, or intolerance of chemoradiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The incidence of weight loss ≥5% during the treatment | From the start to the end of CCRT
  The proportion of patients experiencing a weight loss of 5% or more during the CCRT

SECONDARY OUTCOMES:
Nutrition-related parameters | up to 6 months after radiotherapy
  Nutrition-related parameters, including weight, body mass index (BMI), hemoglobin (HGB), serum albumin (ALB), pre-albumin (PA), lymphocyte (LY)
EORTC Quality of Life Questionnaire C30 (QLQ-C30) | up to 6 months after radiotherapy
  Quality of Life
Scored Patient-Generated Subjective Global Assessment | up to 6 months after radiotherapy
  PG-SGA scores and grades
Toxicities | up to 1 year after radiotherapy
  Treatment-related toxicities, including hematologic adverse effects, radiation pneumonitis, and radiation esophagitis.
Survival outcomes | 3 years
  Including overall survival and progression-free survival.

OTHER OUTCOMES:
Exploratory endpoint | From the start to the end of CCRT
  The association between oral nutritional supplements outcome and the gut microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bovio G, Montagna G, Bariani C, Baiardi P. Upper gastrointestinal symptoms in patients with advanced cancer: relationship to nutritional and performance status. Support Care Cancer. 2009 Oct;17(10):1317-24. doi: 10.1007/s00520-009-0590-x. Epub 2009 Feb 8. PMID 19199106
- [Background] Kiss N, Isenring E, Gough K, Krishnasamy M. The prevalence of weight loss during (chemo)radiotherapy treatment for lung cancer and associated patient- and treatment-related factors. Clin Nutr. 2014 Dec;33(6):1074-80. doi: 10.1016/j.clnu.2013.11.013. Epub 2013 Nov 25. PMID 24325888
- [Background] Unsal D, Mentes B, Akmansu M, Uner A, Oguz M, Pak Y. Evaluation of nutritional status in cancer patients receiving radiotherapy: a prospective study. Am J Clin Oncol. 2006 Apr;29(2):183-8. doi: 10.1097/01.coc.0000198745.94757.ee. PMID 16601440
- [Background] Luo J, Chen YJ, Narsavage GL, Ducatman A. Predictors of survival in patients with non-small cell lung cancer. Oncol Nurs Forum. 2012 Nov;39(6):609-16. doi: 10.1188/12.ONF.609-616. PMID 23107855
- [Background] Sanchez-Lara K, Turcott JG, Juarez E, Guevara P, Nunez-Valencia C, Onate-Ocana LF, Flores D, Arrieta O. Association of nutrition parameters including bioelectrical impedance and systemic inflammatory response with quality of life and prognosis in patients with advanced non-small-cell lung cancer: a prospective study. Nutr Cancer. 2012;64(4):526-34. doi: 10.1080/01635581.2012.668744. Epub 2012 Apr 10. PMID 22489794
- [Background] Ma L, Ye W, Li Q, Wang B, Luo G, Chen Z, Guo S, Qiu B, Liu H. Subjective Global Assessment (SGA) Score Could Be a Predictive Factor for Radiation Pneumonitis in Lung Cancer Patients With Normal Pulmonary Function Treated by Intensity-Modulated Radiation Therapy and Concurrent Chemotherapy. Clin Lung Cancer. 2018 Mar;19(2):e211-e217. doi: 10.1016/j.cllc.2017.09.001. Epub 2017 Sep 19. PMID 29017827
- [Background] Isenring EA, Capra S, Bauer JD. Nutrition intervention is beneficial in oncology outpatients receiving radiotherapy to the gastrointestinal or head and neck area. Br J Cancer. 2004 Aug 2;91(3):447-52. doi: 10.1038/sj.bjc.6601962. PMID 15226773
- [Background] Ravasco P, Monteiro-Grillo I, Marques Vidal P, Camilo ME. Impact of nutrition on outcome: a prospective randomized controlled trial in patients with head and neck cancer undergoing radiotherapy. Head Neck. 2005 Aug;27(8):659-68. doi: 10.1002/hed.20221. PMID 15920748
- [Background] Ravasco P, Monteiro-Grillo I, Vidal PM, Camilo ME. Dietary counseling improves patient outcomes: a prospective, randomized, controlled trial in colorectal cancer patients undergoing radiotherapy. J Clin Oncol. 2005 Mar 1;23(7):1431-8. doi: 10.1200/JCO.2005.02.054. Epub 2005 Jan 31. PMID 15684319
- [Background] Kiss NK, Krishnasamy M, Isenring EA. The effect of nutrition intervention in lung cancer patients undergoing chemotherapy and/or radiotherapy: a systematic review. Nutr Cancer. 2014;66(1):47-56. doi: 10.1080/01635581.2014.847966. Epub 2013 Dec 9. PMID 24320097
- [Background] Sanders KJ, Hendriks LE, Troost EG, Bootsma GP, Houben RM, Schols AM, Dingemans AM. Early Weight Loss during Chemoradiotherapy Has a Detrimental Impact on Outcome in NSCLC. J Thorac Oncol. 2016 Jun;11(6):873-9. doi: 10.1016/j.jtho.2016.02.013. Epub 2016 Mar 3. PMID 26940529